CLINICAL TRIAL: NCT05932550
Title: Safety of Maraviroc for Post-stroke Depression (Proof-of-concept)
Brief Title: Safety of Maraviroc for Post-stroke Depression
Acronym: MRV-PSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0056-20-TLV
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Post-stroke Depression
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Maraviroc 300 mg/day (Experimental): Open-label study
  Interventions: Drug: Maraviroc 300 mg

INTERVENTIONS:
Drug: Maraviroc 300 mg — 10 week treatment as add-on therapy to anti-depressants

SUMMARY:
Post-stroke depression (PSD) is a barrier to effective rehabilitation and recovery after stroke. Current treatment options are limited and there is an unmet need for specific and effective therapeutic options.

Objective: To examine the safety and efficacy of Maraviroc, a CCR5 antagonist, as a possible add-on treatment option for PSD, in an open-labeled proof-of-concept clinical trial.

Design, Setting, and Participants: A 10-week trial of daily oral 300 mg Maraviroc in ten patients with subcortical stroke suffering from PSD. Follow-up: eight weeks after completing treatment.

Main Outcome Measure: A change in the Montgomery-Asberg Depression Rating Scale (MADRS).

ELIGIBILITY:
Inclusion Criteria:

1. 1. Men and women aged 50 to 86 years;
2. Able to fully comprehend and sign an informed consent form;
3. Diagnosis of stroke/TIA prior to study entrance and evidence of ischemic infarct and/or lacunar infarcts on MRI (defined as sharply demarcated hypointense lesions <20mm on T1-weighted images with corresponding hypointense lesions with hyperintense rim on FLAIR) and/or deep Cerebral Microbleeds (CMB) (defined as round hypointense lesions on T2-weighted gradient echo-images with a diameter < 10 mm in neuroimaging.
4. Meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) diagnostic criteria for major depressive episode that developed up to 12 months after the documented stroke/TIA.
5. Able to comply with scheduled visits, treatment plan, and other trial procedures;
6. Treatment with other antidepressants is allowed but subjects will be asked not to change their regular treatment regime during the trial.

   Exclusion Criteria:
7. Hemorrhages and cerebral edema (e.g., subarachnoid haemorrhage, intracerebral hemorrhage, subdural hematoma, epidural hematoma)
8. Patients in a state of coma or with severe disturbance of consciousness, aphasia, agnosia, or deafness that subsequently affects expression and communication.
9. Significant acute medical illness including: drug overdose, severely disturbed liver, kidney or lung function, anemia, hypothyroidism, or uncontrolled diabetes.
10. Significant acute neurologic illness including: impaired consciousness, Parkinson's disease, Huntington's chorea, progressive supranuclear paralysis, brain tumor, subdural hematoma, multiple sclerosis, hydrocephalus, Binswanger's disease, or severe aphasia
11. Patients diagnosed with dementia or major neurocognitive disorder as defined by DSM-5at screening, or other neurological conditions that might dominate the clinical picture (multiple sclerosis, Parkinson's disease, epilepsy, Huntington's chorea, progressive supranuclear paralysis, brain tumor, subdural hematoma, multiple sclerosis, hydrocephalus, Binswanger's disease, etc.)
12. Subject has a history of human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or elevated hepatic transaminases or bilirubin, or tests positive for HIV at Screening.
13. History of renal insufficiency or serum creatinine over 1.6;;
14. Subject has a current or past diagnosis of bipolar or related disorders, intellectual disability, cluster B personality disorder (e.g., borderline personality disorder, antisocial personality disorder, histrionic personality disorder, and narcissistic personality disorder), psychotic disorder, schizophrenia, PTSD , and substance/alcohol use disorders other than nicotine in the past year (including barbiturates, methadone, opiates, cocaine, cannabinoids, and amphetamine/ methamphetamine).
15. Subject has suicidal ideation with intent to act during the screening phase or on Day 1 per investigator's clinical judgment, or has a history of suicidal behavior within the past year; or subject has homicidal ideation/intent at Screening or on Day 1.
16. Subject has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigatoris considered cured with minimal risk of recurrence).
17. Subject has known allergies, hypersensitivity, intolerance, or contraindication to Maraviroc or its excipients.
18. Subject has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 60 days before the planned first dose of study drug or is currently enrolled in an investigational study.
19. Subject is a woman who is pregnant, breast-feeding, or planning to become pregnant while enrolled in this study or within 3 months after the last dose of study drug.
20. Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
21. Subject has had major surgery, (e.g., requiring general anesthesia) within 2 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study.
22. Use of drugs with possible interactions with Maraviroc.

Ages: 50 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 10 weeks
  depression score

SECONDARY OUTCOMES:
16-item quick inventory of depressive symptoms- self-report, QIDS-SR16 | 10 weeks
  self-report depression score
clinical global impression scale (CGI) | 10 weeks
  Clinician impression
7-item patient-reported generalized anxiety disorder 7-item scale- GAD-7 | 10 weeks
  Anxiety score

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data

REFERENCES:
- [Derived] Tene O, Molad J, Rotschild O, Alpernas A, Hawwari M, Seyman E, Giladi N, Hallevi H, Assayag EB. Blocking CCR5 activity by maraviroc augmentation in post-stroke depression: a proof-of-concept clinical trial. BMC Neurol. 2024 Jun 6;24(1):190. doi: 10.1186/s12883-024-03683-3. PMID 38844862